CLINICAL TRIAL: NCT01608295
Title: A Pilot Study of Double-blind Comparison of Vilazodone to Paroxetine in Geriatric Depression
Brief Title: Vilazodone for Treatment of Geriatric Depression
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Principal Investigator, Helen Lavretsky, MD, Professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VII-IT-02
Record Dates: First submitted 2012-05-25; First posted 2012-05-31 (Estimated); Results first posted 2017-05-09 (Actual); Last update posted 2018-05-11 (Actual); Status verified 2018-04

CONDITIONS: Major Depressive Disorder
Keywords: depressed; geriatric; older adults; antidepressants; depression; anxious; major depressive disorder; MDD
MeSH Terms: conditions — Depressive Disorder, Major; Consciousness Disorders; Depression; Anxiety Disorders | interventions — Vilazodone Hydrochloride; Antidepressive Agents; Paroxetine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vilazodone; Viibryd (Experimental): After screening and baseline test results are reviewed and eligibility criteria are confirmed, medications will be dispensed if patients continue to meet eligibility criteria and sign the informed consent form. All eligible subjects will be randomized to vilazodone or paroxetine group using a computer-generated random assignment scheme, which assigned subjects in a 1:1 ratio to each group. Randomization will be done prior to subject's being assigned to the groups. Doses of the drugs will be adjusted according to individual tolerability and safety.
  Interventions: Drug: Vilazodone; Viibryd
- Paroxetine; Paxil (Experimental): After screening and baseline test results are reviewed and eligibility criteria are confirmed, medications will be dispensed if patients continue to meet eligibility criteria and sign the informed consent form. All eligible subjects will be randomized to vilazodone or paroxetine group using a computer-generated random assignment scheme, which assigned subjects in a 1:1 ratio to each group. Randomization will be done prior to subject's being assigned to the groups. Doses of the drugs will be adjusted according to individual tolerability and safety.
  Interventions: Drug: Paroxetine; Paxil

INTERVENTIONS:
Drug: Vilazodone; Viibryd — Subjects randomized to receive vilazodone blindly will have incremental dose titration of 10mg per day for the 1st week; 20mg per day the 2nd week; 40mg per day for the 3rd-12th week. Doses of the drugs will be adjusted according to individual tolerability and safety.
  Other Names: Vilazodone; Viibryd; Antidepressant
  Arms: Vilazodone; Viibryd
Drug: Paroxetine; Paxil — Subjects randomized to receive paroxetine blindly will have incremental dose titration of paroxetine 10mg per day for the 1st week; 20mg per day for the 2nd week; and 30mg per day for the 3rd-12 week. Doses of the drugs will be adjusted according to individual tolerability and safety.
  Other Names: Paroxetine; Paxil; Antidepressant
  Arms: Paroxetine; Paxil

SUMMARY:
The purpose of this study is to examine the effects of vilazodone for the treatment of depression in older adults.

DETAILED DESCRIPTION:
This is a 12-week double-blind comparison of a novel antidepressant, vilazodone, to the gold-standard drug, paroxetine, for the treatment of geriatric depression. We are interested in assessing the difference in response to vilazodone (VLZ) compared to paroxetine (PAR). We hope to detect difference in response in primary outcomes (depressed mood) and secondary outcomes cognition. We are seeking to examine this directly in 80 older adults (60 years of age or older) with major depression with anticipated 60 completers. This proposed trial will serve as a pilot study to estimate the efficacy and tolerability of the drug in older depressed adults, and use this project for dose-finding in this population.

ELIGIBILITY:
Inclusion Criteria:

* 60 years of age or older
* The presence of a major depressive disorder diagnosed according to the Diagnostic and Statistical Manual of Mental Disorders (DSM-IV) criteria
* A 24-item Hamilton Depression Rating Scale (HAMD) score of 17 or higher at baseline
* Mini-Mental State Exam (MMSE) score > 24.

Exclusion Criteria:

* Subjects will be excluded if they had any current and/or lifetime history of other psychiatric disorders (except unipolar depression with or without comorbid generalized anxiety disorder), or recent unstable medical or neurological disorders; any disabilities preventing their participation in the study; diagnosis of mild cognitive impairment (MCI)/dementia; those with known allergic reactions to paroxetine or vilazodone.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2012-07; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Helen Lavretsky, M.D., Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Semel Institute, Los Angeles, California, United States

REFERENCES:
- See also: Double-blind comparison of vilazodone to paroxetine in geriatric depression — http://www.semel.ucla.edu/latelife

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Single site outpatient clinic in the U.S.
Pre-assignment Details: 208 volunteers were assessed for eligibility, of which 100 declined to participate and 37 did not meet inclusion criteria. Seventy-one persons consented to participate, of which 65 passed screening and were enrolled; nine of 65 enrolled participants withdrew before randomization.
Period: Overall Study
Arm/Group | Vilazodone; Viibryd | Paroxetine; Paxil
Started | 26 | 30
Completed | 20 | 25
Not Completed | 6 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vilazodone; Viibryd | Paroxetine; Paxil | Total
Number analyzed (Participants) | 26 | 30 | 56
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 9 | 14
  >=65 years | 21 | 21 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.5 (7.2) | 71.5 (7.7) | 71.5 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 13 | 26
  Male | 13 | 17 | 30
Region of Enrollment [Number; unit: participants]
  United States | 26 | 30 | 56

OUTCOME MEASURES:

1. Primary Outcome: Hamilton Depression Rating Scale (HDRS)
Description: The HAMD measures the severity of depressive symptoms in participants with major depressive disorder (MDD). It is a checklist of 17 items that are ranked on a scale of 0-4 or 0-2. The range for the total score (which is the sum of the scores of all 17 items) is 0-52; a higher score indicates greater severity of symptoms.
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Vilazodone; Viibryd: Vilazodone; Viibryd: Subjects randomized to receive vilazodone blindly received incremental dose titration of 10mg per day for the 1st week; 20mg per day the 2nd week; 40mg per day for the 3rd-12th week. Doses of the drugs will be adjusted according to individual tolerability and safety.
- Paroxetine; Paxil: Paroxetine; Paxil: Subjects randomized to receive paroxetine blindly received incremental dose titration of paroxetine 10mg per day for the 1st week; 20mg per day for the 2nd week; and 30mg per day for the 3rd-12 week. Doses of the drugs were adjusted according to individual tolerability and safety.
Arm/Group | Vilazodone; Viibryd | Paroxetine; Paxil
Number analyzed (Participants) | 21 | 25
units on a scale
  HDRS Baseline | 17.2 (3.7) | 16.6 (4.1)
  HDRS Final Visit | 7.6 (4.8) | 7.5 (5.9)

2. Secondary Outcome: UKU Side-effect Profile
Description: Number of participants with each side-effect event.
Time Frame: Each visit for 12 weeks
Measure: Number; unit: participants
Arm/Group | Vilazodone; Viibryd | Paroxetine; Paxil
Number analyzed (Participants) | 25 | 30
participants
  Concentration Difficulties | 3 | 0
  Sedation | 1 | 3
  Increased dream activity | 3 | 3
  Reduced salivation | 3 | 1
  Diarrhea | 3 | 1
  Constipation | 3 | 5
  Orthostatic dizziness | 3 | 3

3. Secondary Outcome: Neurocognitive Measure: The Rey-Osterrieth Complex Figure Test
Description: The The Rey-Osterrieth Complex Figure Test (REY-O) is a neuropsychological assessment in which measures visual perception and long-term visual memory. Total raw scores range from 0 to 36 with higher scores representing better outcomes in recall. The total raw score represents a sum of subscales scored by 18 individual elements which are scored for both distortion and placement. Two points are awarded to elements that are accurately drawn and properly placed, one point is given to distorted or misplaced elements, 0.5 points are given if an element is both distorted and misplaced, and missing or unrecognizable elements receive zero points.
Time Frame: Baseline and Final Visit
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Vilazodone; Viibryd | Paroxetine; Paxil
Number analyzed (Participants) | 20 | 25
units on a scale
  REY-O 3 Minute Delay Baseline | 13.3 (5.9) | 13.3 (5.3)
  REY-O 3 Minute Delay Final Visit | 15.2 (7.4) | 16.3 (4.8)

4. Secondary Outcome: Changes in Proinflammatory Gene Expression From Baseline to Final Visit (up to 12 Weeks)
Description: Gene expression data were quantile-normalized and log2-transformed in RNA expression units. The measure included the promoter transcription factor binding motif prevalence ratio of the unit (log2 Vilazodone/Paroxetine) and ranging from a minimum of -3 to a maximum of 3 with higher scores indicating better outcomes.
Time Frame: Baseline and Final Visit
Population: The Arms/Groups are not combined, but results are presented as a ratio of Vilazodone/Paroxetine.
Measure: Mean (Standard Error); unit: RNA expression units
Groups:
- Vilazodone and Paroxetine: Subjects randomized to receive vilazodone relative to subjects randomized to receive paroxetine.
Arm/Group | Vilazodone and Paroxetine
Number analyzed (Participants) | 46
RNA expression units
  AP-1, Activator Protein | -0.8 (0.5)
  NF-kB, Nuclear Factor Kappa B | -1.25 (0.5)
  GR, Glucocorticoid Receptor | 0.2 (0.6)
  CREB, cAMP response element binding protein | -2.1 (0.7)

ADVERSE EVENTS:
Arm/Group | Vilazodone; Viibryd | Paroxetine; Paxil
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/30
Other Adverse Events (participants affected / at risk) | 19/26 | 16/30
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vilazodone; Viibryd (N=26) | Paroxetine; Paxil (N=30)
Reduced salivation (Gastrointestinal disorders) | 3 | 1
Concentration Difficulties (Psychiatric disorders) | 3 | 0
Sedation (Nervous system disorders) | 1 | 3
Increased Dream Activity (Nervous system disorders) | 3 | 3
Diarrhea (Gastrointestinal disorders) | 3 | 1
Constipation (Gastrointestinal disorders) | 3 | 5
Orthostatic dizziness (Vascular disorders) | 3 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No